CLINICAL TRIAL: NCT00576082
Title: DIVERSITY OF BORRELIA SPECIES INVOLVED IN CUTANEOUS MANIFESTATIONS OF LYME BORRELIOSIS IN FRANCE
Brief Title: Borrelia Species in Cutaneous Lyme Borreliosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Other Study IDs: 3977
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Lyme Borreliosis
Keywords: Lyme borreliosis; Erythema migrans; Borrelial lymphocytoma; Acrodermatitis chronica atrophicans; Borrelia burgdorferi; Borrelia afzelii; Borrelia garinii
MeSH Terms: conditions — Lyme Disease; Glossitis, Benign Migratory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cutaneous biopsy specimen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cutaneous biopsy — Cutaneous biopsy in order to search Borrelia by means of culture and PCR in this tissue sample

SUMMARY:
The aim of this study is to identify the species of Borrelia involved in the dermatologic manifestations of Lyme borreliosis in France. Indeed, in Europe, as opposed to North America, many bacterial species are involved in Lyme borreliosis. Yet, very few is known about the prevalence and distribution of different bacteriological species that account for the disease in France. Thus, this a nation-wide study in which all French dermatologists are invited to participate. Every adult patient presenting with one of the cutaneous manifestation of Lyme borreliosis: erythema migrans, lymphocytoma or acrodermatitis chronica atrophicans can be included in the study. If the patient agrees participating, after information and written consent, a cutaneous biopsy will be performed in order to isolate Borrelia by means of culture and PCR. An estimated 400 biopsies should be performed within 2 years.

ELIGIBILITY:
Inclusion criteria:

* Informed adult patient who signed written consent with one the following conditions:
* erythema migrans
* borrelial lymphocytoma
* acrodermatitis chronica atrophicans

Exclusion criteria:

* pregnancy or lactation
* allergy to local anesthesia
* patient who refuses biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every adult patient presenting with either erythema migrans, borrelial lymphocytoma or acrodermatitis chronica atrophicans
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2008-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dan LISPKER, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Service de Dermatologie, Hôpital Civil, Strasbourg
  - Service des Maladies infectieuses et tropicales, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg